CLINICAL TRIAL: NCT02966990
Title: Biomechanical Analysis of the Effects of Upper Limb Orthosis During the Execution of a Functional Task
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Flavia Pessoni Faleiros Macedo Ricci, PhD Student, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPGRDF-FMRP-USP
Record Dates: First submitted 2016-11-07; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Orthotic Devices; Electromyography; Biomechanical Phenomena; Hand; Upper Extremity Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hand orthosis patients (Other): Patients using hand orthosis for better hand function
  Interventions: Device: Hand Orthotic Devices

INTERVENTIONS:
Device: Hand Orthotic Devices — Orthotic device made to provide the patient with better hand function

SUMMARY:
The orthotics are auxiliary therapeutic resources indicated for the relief of pain, improves functional standard or correction of deformities. There is a lack of studies that analyze the biomechanical changes promoted by the Orthotics in functional pattern of the upper limb. The objective of this proposal is to analyse biomechanical changes in the functional upper limb pattern with the use of orthoses for patients with dysfunctions arising from musculoskeletal system trauma or burns, aiming to contribute with scientific evidence to clinical practice. The project will analyze the changes in the pattern of the upper limb functional through the use of dynamic and static Orthotics by means of kinematic and electromyographic analysis while conducting a functional task. These comparisons will be carried out with and without the use of functional Orthotics, and the controls are the patients themselves. Methods: 25 patients will be included over 18 years with malfunctions resulting from orthopaedic trauma and Burns of the upper limb with indication and Orthotics for improving functional pattern. For characterization of the sample will be performed: esthesiometric , hand and the (Disabilities of the Arm, Shoulder and Hand) DASH Questionnaire. Biomechanical assessment will be used for the analysis and electromyographic kinematics. For statistical analysis will be applied the method of analysis of variance (ANOVA) for repeated measures, and when necessary, the post hoc Bonferroni test. Will be adopted as significance level p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients who are using hand orthosis for functional purposes

Exclusion Criteria:

* neurological problems; cognitive deficits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Electromyographic assessment | one day
  Muscle activity will be measured using surface EMG (TrignoTM Wireless System, Delsys, USA), collected at a sample rate of 2000 Hz.
Kinematic analysis | one day
  Movements will be recorded with a ViconTM (Oxford Metrics, UK) motion capture eight-camera system operating at a frequency of 200 Hz.

SECONDARY OUTCOMES:
Functional assessment | one day
  The DASH questionnaire will be applied and Grip strength will be measured

IPD SHARING:
Plan to Share IPD: No